CLINICAL TRIAL: NCT06206057
Title: The Relationship Between Leisure Activities and Aging Anxiety in Middle-aged Women
Brief Title: The Relationship Between Leisure Activities and Aging Anxiety in Women
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Buğu Usanma Koban, Asst Prof in Family Medicine Department, Marmara University Pendik Training and Research Hospital
Other Study IDs: 09.2023.1457
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Aging; Anxiety; Premenopause; Womans Health
Keywords: aging; women's health; anxiety; leisure activities
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the effect of leisure activities on aging anxiety of middle-aged (45-59) women. The main question it aims to answer is: Do the leisure activities (doing sports, playing music instruments, doing handicrafts, writing, taking care of a pet, growing plants, dancing etc.) affect the aging anxiety level of middle-aged women? Participants will be required to fill out a form querying their socio-demographic information, medical histories, and regular leisure activities. Subsequently, the "Aging Anxiety Scale for Middle-Aged Women" will be applied.

DETAILED DESCRIPTION:
In this study, women aged between 40 and 59 registered at the Marmara University Education Family Health Center (FHC) in the Tuzla district will be included. There are a total of 352 women in this age range registered with the FHC, and it is aimed to reach all of them.

Patients will be informed about the study by Dr. Buğu Usanma Koban via telephone, and they will be invited to the FHC for the administration of the questionnaire. After obtaining informed consent from those who agree to participate in the study, their personal information will be recorded through a face-to-face interview. Subsequently, the Aging Anxiety Scale for Middle-Aged Women, developed by Lee and You, and validated in Turkish by Aydın and Kabasakal, will be applied to the participants.

Finally, volunteers will be asked to fill out a questionnaire specifying the types and frequencies of their leisure activities. SPSS (version 20.0, SPSS Inc., Chicago, IL, USA) will be used for data analysis.

Descriptive statistical information will be presented as mean ± standard deviation or %, and a p-value less than 0.05 will be considered statistically significant. In the comparison of more than two independent groups that do not meet the assumptions of parametric tests, the Kruskal-Wallis analysis will be conducted. If the analysis is significant, groups will be subjected to pairwise Mann-Whitney U tests.

To understand the relationship between leisure activities and aging anxiety, Spearman Correlation Analysis will be conducted for parameters conforming to normal distribution, and Pearson Correlation Analysis will be performed for parameters not conforming to normal distribution. The correlation coefficient (r value) will be specified.

ELIGIBILITY:
Inclusion Criteria:

* Not having a medical condition that requires urgent intervention or hospitalization
* Not having psychological or physical barrier preventing communication.

Exclusion Criteria:

* a medical condition that requires urgent intervention or hospitalization
* having a psychological or physical barrier preventing communication.

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged between 40 and 59 registered at the Marmara University Education Family Health Center (FHC) in the Tuzla district
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Effect of leisure activities on aging anxiety | 3 months
  Relationship between leisure activities' type and frequency, and scores of Aging Anxiety Scale for Middle-Aged Women will be investigated.
  The scale consists of 19 questions and is scored on a 5-point Likert scale. The highest possible score on the scale is 95, and the lowest score is 19. Obtaining a high score indicates a high level of aging anxiety.

SECONDARY OUTCOMES:
Sociodemographic properties and aging anxiety | 3 months
  In the form created for collecting sociodemographic information, marital status (married, single, widowed/divorced) and educational status (illiterate, literate, primary school graduate, high school graduate, university and college graduate) will be queried. The correlation between the answers and the scores on the "Aging Anxiety Scale for Middle-Aged Women" will be examined.
  The scale consists of 19 questions and is scored on a 5-point Likert scale. The highest possible score on the scale is 95, and the lowest score is 19. Obtaining a high score indicates a high level of aging anxiety.
Effect of chronic diseases on aging anxiety | 3 months
  Correlation between number and type of chronic diseases and the scores on the "Aging Anxiety Scale for Middle-Aged Women" will be examined.
  The scale consists of 19 questions and is scored on a 5-point Likert scale. The highest possible score on the scale is 95, and the lowest score is 19. Obtaining a high score indicates a high level of aging anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Buğu Usanma Koban, Asst Dr, Principal Investigator — Marmara University Medical School
Locations (1):
- Marmara University Education Family Healthcare Center, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barrett AE, Robbins C. The multiple sources of women's aging anxiety and their relationship with psychological distress. J Aging Health. 2008 Feb;20(1):32-65. doi: 10.1177/0898264307309932. Epub 2007 Dec 18. PMID 18089765
- [Background] Barrett AE, Toothman EL. Multiple "Old Ages": The Influence of Social Context on Women's Aging Anxiety. J Gerontol B Psychol Sci Soc Sci. 2018 Oct 10;73(8):e154-e164. doi: 10.1093/geronb/gbx027. PMID 28453655
- [Background] Oh A, Kim J, Yi E, Shin J. Verification of the Mediating Effect of Social Support on Physical Activity and Aging Anxiety of Korean Pre-Older Adults. Int J Environ Res Public Health. 2020 Nov 2;17(21):8069. doi: 10.3390/ijerph17218069. PMID 33147775